CLINICAL TRIAL: NCT03435523
Title: Optimal PEEP Based on the Open Lung Approach During One Lung Ventilation in Thoracic Surgery: a Physiological Study.
Brief Title: The Open Lung Approach During One Lung Ventilation in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Gilda Cinnella, Associate Professor, University of Foggia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Università di Foggia
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open lung approach (Experimental): Recruitment maneuver during OLV in thoracic surgery
  Interventions: Procedure: Recruitment maneuver

INTERVENTIONS:
Procedure: Recruitment maneuver — the ventilator was switched to pressure-control ventilation with a driving pressure of 20 cmH2O. After a 3 min equilibration, PEEP was applied in steps of 5,10,15 and 20 cmH2O every five respiratory breaths; subsequently, after setting a driving pressure of 15 cmH2O, PEEP was stepwise reduced, starting from 15 cmH2O, by 2 cmH2O every 2 minutes. The recruiting pressure of 20/20 was applied for six breaths. During the decremental PEEP trial, CRS was measured at every step. The PEEP level corresponding to highest CRS during the decremental trial was identified as the "best PEEP". Subsequently, the lungs were recruited again and the "best" PEEP was applied.

SUMMARY:
* Question: Ventilatory strategy to counterbalance the effect of one lung ventilation during thoracic surgery.
* Findings: the open lung approach improved oxygenation and lung compliance, reducing respiratory system driving pressure and transpulmonary driving pressure.
* Meaning: patients undergoing thoracic surgery during one lung ventilation may benefit of an open lung approach strategy to avoid ventilator lung injury.

DETAILED DESCRIPTION:
Background: During thoracic surgery in lateral decubitus, one lung ventilation (OLV) may impair respiratory mechanics and gas exchange. The investigators tested a strategy based on an open lung approach (OLA) consisting in lung recruitment immediately followed by a decremental positive-end expiratory pressure (PEEP) titration to the best respiratory system compliance (CRS) and separately quantified the elastic properties of the lung and the chest wall. The investigators hypothesis was that this approach would improve gas exchange and increase lung compliance (CL).

Methods: In thirteen patients undergoing upper left lobectomy the investigators studied lung and chest wall mechanics, transpulmonary pressure (PL), respiratory system and transpulmonary driving pressure (ΔPRS and ΔPL), gas exchange and hemodynamics at two time-points (a) during OLV at zero end-expiratory pressure (OLVpre-OLA) and (b) after the application of the open-lung strategy (OLVpost-OLA).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* surgery and OLV lasting ≥ 60 min

Exclusion Criteria:

* lung reduction surgery, pneumonectomy, patients with severe COPD with preoperative forced expiratory volume in 1 s (FEV1) to forced vital capacity (FVC) ratio, expressed as a percentage (FEV1/FVC%) <60%, presence of large bullae, pleural diseases and/or acute or chronic uncompensated cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Change in respiratory mechanics before and after the open lung approach | During surgery
  Respiratory mechanics parameters were recorded, digitized and collected on a personal computer through a 12-bit analog-to digital converter board (DAQCard 700; National Instrument, Austin, TX) at a sample rate of 200 Hz (ICU Lab, KleisTEK Engineering, Bari, Italy).

REFERENCES:
- [Derived] Rauseo M, Mirabella L, Grasso S, Cotoia A, Spadaro S, D'Antini D, Valentino F, Tullo L, Loizzi D, Sollitto F, Cinnella G. Peep titration based on the open lung approach during one lung ventilation in thoracic surgery: a physiological study. BMC Anesthesiol. 2018 Oct 31;18(1):156. doi: 10.1186/s12871-018-0624-3. PMID 30382819